CLINICAL TRIAL: NCT01300468
Title: A Phase I Study of Oral PHA-848125AC Given Daily For 7 Consecutive Days Every 2 Weeks or for 4 Consecutive Days A Week for 3 Consecutive Weeks Every 4 Weeks to Adult Patients With Advanced/Metastatic Solid Tumors
Brief Title: Study of PHA-848125AC in Adult Patients With Advanced/Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Clinical Research Head, Nerviano Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDKO-125a-001
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Solid Tumour
Keywords: advanced/metastatic solid tumors
MeSH Terms: interventions — N,1,4,4-tetramethyl-8-((4-(4-methylpiperazin-1-yl)phenyl)amino)-4,5-dihydro-1H-pyrazolo(4,3-h)quinazoline-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose-escalation (Experimental)
  Interventions: Drug: PHA-848125AC

INTERVENTIONS:
Drug: PHA-848125AC

SUMMARY:
The purpose of this open-label, multi center, Phase I study was to determine the safety profile of the oral compound PHA-848125AC administered according to two different schedules of administrations to advanced/metastatic solid tumor patients. Objectives of the study were to determine the maximum tolerated dose and the dose that can be recommended for Phase II investigations.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written IRB-approved Informed Consent
* Histologically or cytologically confirmed relapsed or refractory solid tumors for which no standard therapy exists
* ECOG (WHO) performance status 0-1
* Life expectancy of at least 3 months
* Age >=18 years
* A negative pregnancy test (if female in reproductive years)
* Acceptable liver and renal function
* Acceptable hematologic status
* 10. Previous cancer therapy is allowed with the exclusion of experimental CDK2 inhibitors. Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy must be completed within one month prior to study entry
* Use of effective contraceptive methods if men and women of child producing potential
* Capability to swallow capsules intact
* Grade <=1 retinopathy

Exclusion Criteria:

* In the past 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
* Known brain metastases
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or breast feeding women
* Unwillingness or inability to comply with procedures required in this protocol
* Known infection with HIV, active hepatitis B or hepatitis C
* Diabetes mellitus uncontrolled, or with clinical evidence of diabetic retinopathy, severe peripheral vascular disease or diabetic ulcers
* Current enrollment in another clinical trial
* Patients who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation (lactose intolerance)
* Previous history or current presence of neurological disorders, including epilepsy (although controlled by anticonvulsant therapy), Parkinson's disease, multiple sclerosis, stroke and cerebellar injury
* Gastrointestinal disease (e.g. Crohn's disease, ulcerative colitis, or short gut syndrome) that would impact on drug absorption
* Chronic/intensive use of antacid or H2 receptor antagonists
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the investigator and/or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determination of Dose Limiting Toxicities and Maximum Tolerated Dose | First cycle

SECONDARY OUTCOMES:
Assessment of Adverse Events (based on CTCAE version 3.0) | All cycles
Evaluation of pharmacokinetics: plasma concentrations at different times after dosing and related assessment of conventional pharmacokinetic parameters | First 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Von Hoff, MD, Principal Investigator — Scottsdale Clinical Research Institute, Scottsdale AZ, USA; Manuel Hidalgo, MD, Principal Investigator — The Johns Hopkins University, Baltimore MD, USA; Daniel Laheru, MD, Principal Investigator — The Johns Hopkins University, Baltimore MD, USA
Locations (2):
- United States (2):
  - Scottsdale Clinical Research Institute, Scottsdale, Arizona
  - The Johns Hopkins University, Baltiomore, Maryland